CLINICAL TRIAL: NCT01446146
Title: Increasing Engagement in PTSD Treatment Through Patient Education and Patient Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: South Central VA Mental Illness Research, Education & Clinical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Juliette Mott, Principal Investigator, Michael E. DeBakey VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-28111
Record Dates: First submitted 2011-09-28; First posted 2011-10-05 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Posttraumatic Stress Disorder; PTSD Treatment; Decision making; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

ARMS (2):
- IDM intervention (Experimental): Will receive a 40 minute intervention session with a clinician, learning about PTSD treatment options and choosing a preferred treatment.
  Interventions: Behavioral: Informed decision making
- Treatment as usual plus placebo session (Placebo Comparator): Will work with provider to select a treatment plan and will receive a 40 minute session without IDM intervention.
  Interventions: Behavioral: Placebo session

INTERVENTIONS:
Behavioral: Informed decision making — 40 minute session with a clinician. Participants will learn about the available PTSD treatment options and will be given a decision aid with more information.
  Arms: IDM intervention
Behavioral: Placebo session — Participant will complete clinician-administered measures in a 40-minute session.
  Arms: Treatment as usual plus placebo session

SUMMARY:
The purpose of this program is to compare two different methods of matching a Veteran to a PTSD treatment.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD) is a serious disorder that affects many Veterans who have had a traumatic experience. The VA offers several different types of treatment for PTSD. We are researching different ways to match a Veteran to a type of treatment. Participants in this study will will be randomly assigned to either a 40-minute session in which they will learn about PTSD treatments and select a preferred treatment or to a 40-minute assessment interview. Those participants assigned to the assessment interview will have the opportunity to work with their Trauma Recovery Program provider to determine a plan for their PTSD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of combat-related PTSD
* Newly enrolled in Trauma Recovery Program (TRP) at the Michael E. DeBakey VA medical center
* TRP provider approval

Exclusion Criteria:

* Previous participation in TRP treatment for PTSD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Treatment participation | 4 months
  Trauma Recovery Program service utilization as assessed by chart review.

SECONDARY OUTCOMES:
Treatment satisfaction | 4 months
  Assessed via self-report measures (Client Satisfaction Questionnaire, Credibility/Expectancy Questionnaire) and semi-structured interview
Change in PTSD severity | Baseline and 4 months
  Assessed by the PCL-M at baseline and 4 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Juliette M Mott, PhD, Principal Investigator — MDVAMC, BCM, SC MIRECC
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States